CLINICAL TRIAL: NCT02190747
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Efficacy and Safety Study of a RARγ-Specific Agonist (Palovarotene) in the Treatment of Preosseous Flare-ups in Subjects With Fibrodysplasia Ossificans Progressiva (FOP)
Brief Title: An Efficacy and Safety Study of Palovarotene to Treat Preosseous Flare-ups in FOP Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clementia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PVO-1A-201; 2014-001453-17 (EudraCT Number)
Record Dates: First submitted 2014-07-13; First posted 2014-07-15 (Estimated); Results first posted 2020-06-24 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Fibrodysplasia Ossificans Progressiva
Keywords: Intervention study; Clinical trial Phase 2; Efficacy and safety; Heterotopic ossification; Flare-up; Palovarotene; Retinoic acid receptor agonist; Retinoic acid receptor gamma agonist; Clementia; Myositis Ossificans Progressiva; Munchmeyer's Disease; FOP
MeSH Terms: conditions — Myositis Ossificans; Ossification, Heterotopic | interventions — Palovarotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Palovarotene dose level 1 (Cohort 1) (Experimental): Doses of palovarotene in dose level 1 are 10 mg once daily for 14 days, followed by 5 mg once daily for 28 days.
  Interventions: Drug: Palovarotene
- Palovarotene dose level 2 (Cohort 2) (Experimental): Weight-adjusted doses of palovarotene in dose level 2 are 10 mg palovarotene once daily, followed by 5 mg once daily for 28 days.
  Interventions: Drug: Palovarotene
- Palovarotene dose level 3 (Cohort 2) (Experimental): Weight-adjusted doses of palovarotene in dose level 3 are 5 mg palovarotene once daily, followed by 2.5 mg once daily for 28 days.
  Interventions: Drug: Palovarotene
- Sugar pill (Placebo Comparator): The placebo comparator will be taken once daily for the same duration as the palovarotene dose groups in both Cohorts 1 and 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Palovarotene — Palovarotene will be taken orally once daily at approximately the same time each day. Powder filled hard gelatin capsules will be opened and the contents added onto specific food.
  Arms: Palovarotene dose level 1 (Cohort 1); Palovarotene dose level 2 (Cohort 2); Palovarotene dose level 3 (Cohort 2)
Drug: Placebo
  Arms: Sugar pill

SUMMARY:
Fibrodysplasia ossificans progressiva (FOP) is a rare, severely disabling disease characterized by painful, recurrent episodes of soft tissue swelling (flare-ups) that result in abnormal bone formation in muscles, tendons, and ligaments. Flare-ups begin early in life and may occur spontaneously or after soft tissue trauma, vaccinations, or influenza infections. Recurrent flare-ups progressively restrict movement by locking joints leading to cumulative loss of function and disability. Mouse models of FOP have demonstrated the ability of retinoic acid receptor (RAR) gamma agonists to prevent heterotopic ossification (HO) following injury. The purpose of the study is to evaluate whether palovarotene, an RAR gamma agonist, will prevent HO during and following a flare-up in subjects with FOP.

DETAILED DESCRIPTION:
The primary objective is to evaluate the ability of different doses of palovarotene to prevent HO at the flare-up site in subjects with FOP as assessed by plain radiographs.

This is a Phase 2, multi-center, randomized, double-blind, sponsor-unblinded, placebo-controlled study. Two cohorts of subjects will be randomized into different dosing regimens of palovarotene for a 6-week (42 days) treatment period. The study will consist of three periods:

1. A Screening period to occur within 7 days of a distinct flare-up. The first dose of study drug will be taken within 7 days of the flare-up initiation.
2. A double-blind treatment period of 6 weeks (42 days) duration.
3. A follow-up period of 6 weeks (42 days) duration.

An initial cohort (Cohort 1) of subjects will be randomly assigned 3:1 to either palovarotene or placebo daily for 42 days. Subjects randomized to palovarotene in Cohort 1 will receive an initial daily dose of 10 mg for 14 days followed by 5 mg daily for 28 days.

In Cohort 2, new FOP subjects meeting all inclusion/exclusion criteria will be randomly assigned 3:3:2 to two dose regimens of palovarotene (10 mg for 14 days and 5 mg for 28 days; 5 mg for 14 days and 2.5 mg for 28 days) or placebo daily for 42 days. Doses will be weight-adjusted and subjects randomized within three weight-range categories (20 to <40 kg, 40 to <60 kg, and ≥60 kg).

Subjects completing the study and still meeting eligibility requirements will be given the opportunity to enroll into an open-label extension study.

ELIGIBILITY:
Inclusion Criteria:

* Written, signed, and dated informed subject/parent consent or age-appropriate assent.
* Subjects clinically diagnosed with classic Fibrodysplasia Ossificans Progressiva (FOP).
* Symptomatic onset of a distinct flare-up within 7 days of Study Day 1 (start of study drug) and defined by the presence of at least two of six of the following symptoms: pain, soft tissue swelling, decreased range of motion, stiffness, redness, and warmth. Flare-up must be confirmed by the physician at the Screening visit.
* Flare-up is at an appendicular area (upper or lower extremity), abdomen, or chest; and subject has received, is receiving, or is willing to receive treatment per standard of care, which may or may not include oral prednisone (2 mg/kg PO to a maximum dose of 100 mg daily) for 4 days.
* Abstinent or using two highly effective forms of birth control.
* Subjects must be accessible for treatment and follow-up. Subjects living at distant locations from the investigational site must be able and willing to travel to a site for the initial and all follow-up visits.

Exclusion Criteria:

* Weight <20 kg.
* Intercurrent non-healed fracture at any location.
* Complete immobilization of joint at site of flare-up.
* The inability of the subject to undergo imaging assessments using plain radiographs.
* If currently using vitamin A or beta carotene, multivitamins containing vitamin A or beta carotene, or herbal preparations, fish oil, and unable or unwilling to discontinue use of these products for the duration of the study.
* Exposure to synthetic oral retinoids in the past 30 days prior to Screening (signature of the informed consent).
* Concurrent treatment with tetracycline due to the potential increased risk of pseudotumor cerebri.
* History of allergy or hypersensitivity to retinoids or lactose.
* Concomitant medications that are inhibitors or inducers of CYP450 3A4 activity.
* Amylase or lipase >1.5x above the upper limit of normal or with a history of chronic pancreatitis.
* Elevated aspartate aminotransferase or alanine aminotransferase >2.5x the upper limit of normal.
* Fasting triglycerides >400 mg/dL with or without therapy.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07-14 (Actual); Primary Completion 2016-05-23 (Actual); Study Completion 2016-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (4):
- United States (2):
  - University of California San Francisco, Division of Endocrinology and Metabolism, San Francisco, California
  - University of Pennsylvania, Center for Research in FOP & Related Disorders, Philadelphia, Pennsylvania
- Hôpital Necker-Enfants Malades, Department of Genetics, Paris, France
- The Royal National Orthopaedic Hospital, Brockley Hill, Stanmore, Middlesex, United Kingdom

REFERENCES:
- [Background] Shimono K, Tung WE, Macolino C, Chi AH, Didizian JH, Mundy C, Chandraratna RA, Mishina Y, Enomoto-Iwamoto M, Pacifici M, Iwamoto M. Potent inhibition of heterotopic ossification by nuclear retinoic acid receptor-gamma agonists. Nat Med. 2011 Apr;17(4):454-60. doi: 10.1038/nm.2334. Epub 2011 Apr 3. PMID 21460849
- [Derived] Pignolo RJ, Al Mukaddam M, Baujat G, Brown MA, De Cunto C, Hsiao EC, Keen R, Le Quan Sang KH, Grogan DR, Marino R, Strahs AR, Kaplan FS. Study methodology and insights from the palovarotene clinical development program in fibrodysplasia ossificans progressiva. BMC Med Res Methodol. 2023 Nov 13;23(1):269. doi: 10.1186/s12874-023-02080-7. PMID 37957586
- [Derived] Lindborg CM, Al Mukaddam M, Baujat G, Cho TJ, De Cunto CL, Delai PLR, Eekhoff EMW, Haga N, Hsiao EC, Morhart R, de Ruiter R, Scott C, Seemann P, Szczepanek M, Tabarkiewicz J, Pignolo RJ, Kaplan FS. Most Fractures Treated Nonoperatively in Individuals With Fibrodysplasia Ossificans Progressiva Heal With a Paucity of Flareups, Heterotopic Ossification, and Loss of Mobility. Clin Orthop Relat Res. 2023 Dec 1;481(12):2447-2458. doi: 10.1097/CORR.0000000000002672. Epub 2023 May 8. PMID 37156007
- [Derived] Pignolo RJ, Kimel M, Whalen J, Kawata AK, Artyomenko A, Kaplan FS. The Fibrodysplasia Ossificans Progressiva Physical Function Questionnaire (FOP-PFQ): A patient-reported, disease-specific measure. Bone. 2023 Mar;168:116642. doi: 10.1016/j.bone.2022.116642. Epub 2022 Dec 13. PMID 36526263
- [Derived] Pignolo RJ, Baujat G, Hsiao EC, Keen R, Wilson A, Packman J, Strahs AL, Grogan DR, Kaplan FS. Palovarotene for Fibrodysplasia Ossificans Progressiva (FOP): Results of a Randomized, Placebo-Controlled, Double-Blind Phase 2 Trial. J Bone Miner Res. 2022 Oct;37(10):1891-1902. doi: 10.1002/jbmr.4655. Epub 2022 Aug 17. PMID 35854638
- See also: Website for the International FOP Association — http://ifopa.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight subjects were randomized 3:1 to either palovarotene or placebo in Cohort 1; 8 additional subjects were randomized 3:1 in an interim period between Cohorts 1 and 2. In Cohort 2, 24 additional fibrodysplasia ossificans progressiva (FOP) subjects were randomized 3:3:2 across 2 weight-based regimens of palovarotene or placebo.
Pre-assignment Details: The study included clinically diagnosed FOP subjects at least 6 years of age (Cohort 2) or 15 years of age and older (Cohort 1) with symptomatic onset of a flare-up within 7 days of treatment start and accessible for treatment and follow-up.
Groups:
- Palovarotene 10/5 mg: Subjects received palovarotene 10 milligram (mg) orally for 14 days followed by 5 mg orally for 28 days during flare-ups (10/5 mg regimen). The subjects were followed for an additional 42 days without treatment. Subjects in Cohort 1 and Cohort 2 contributed to this arm.
- Palovarotene 5/2.5 mg: Subjects received palovarotene 5 mg orally for 14 days followed by 2.5 mg orally for 28 days during flare-ups (5/2.5 mg regimen). The subjects were followed for an additional 42 days without treatment. Only subjects in Cohort 2 contributed to this arm.
- Placebo: Subjects received placebo (matching with palovarotene) for 42 days during flare-ups. Subjects were followed for an additional 42 days without treatment. Subjects in Cohort 1 and Cohort 2 contributed to this arm.
Period: Overall Study
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg | Placebo
Started | 21 | 9 | 10
Completed | 21 | 9 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all subjects who received at least 1 dose of study drug (placebo or palovarotene).
Groups:
- Palovarotene 10/5 mg: Subjects received palovarotene 10 mg orally for 14 days followed by 5 mg orally for 28 days during flare-ups (10/5 mg regimen). The subjects were followed for an additional 42 days without treatment. Subjects in Cohort 1 and Cohort 2 contributed to this arm.
- Total: Total of all reporting groups
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg | Placebo | Total
Number analyzed (Participants) | 21 | 9 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.8 (10.3) | 17.9 (8.6) | 21.2 (13.7) | 21.3 (10.8)
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 3 | 4 | 2 | 9
  Adolescents (12-17 years) | 5 | 0 | 4 | 9
  Adults (18-64 years) | 13 | 5 | 4 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 7 | 22
  Male | 12 | 3 | 3 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 13 | 8 | 6 | 27
  Unknown or Not Reported | 6 | 0 | 3 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 7 | 6 | 25
  Black or African American | 1 | 1 | 0 | 2
  Asian | 0 | 0 | 1 | 1
  Multiple | 2 | 1 | 0 | 3
  Not available | 6 | 0 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders at Week 6
Description: A responder was defined as a subject with no or minimal new heterotopic ossification (HO) at flare-up site versus baseline as assessed by plain radiographs at Week 6. Minimal new HO is defined as new HO with an HO score <=3 in both anterior/posterior (AP) and lateral projections (or if one view is non-interpretable or non-evaluable, then remaining evaluable view is used). The HO score ranges from 0 to 6 where, 0 = no HO and 6 = single contiguous HO with longest dimension >2 diameters of reference normotopic bone in any projection. The highest HO score from the 2 projections was used. Results from Primary Read reviews are presented. The Primary Read process included a double-read radiology review paradigm with consensus adjudication. Radiography and CT scans were examined independently by scan type, flare-up region, and imaging time point in order to determine whether radiography would be sufficient to measure new HO formation. Only subjects with interpretable outcomes were evaluated.
Time Frame: Baseline (Day 1) and Week 6 (Day 42)
Population: The Per Protocol (PP) population included all subjects who were eligible for full analysis set (FAS) population, completed Week 6 study visit with no major protocol deviations with at least 80% compliance with study drug, and had an evaluable radiograph or computed tomography (CT) at Week 6 sufficient to allow determination of HO at flare-up site.
Measure: Number; unit: percentage of subjects
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg | Placebo
Number analyzed (Participants) | 20 | 9 | 9
percentage of subjects | 100 | 88.9 | 88.9
Statistical Analysis 1: Comparison: Palovarotene 10/5 mg vs Palovarotene 5/2.5 mg vs Placebo; Cochran-Armitage test of trend (one-sided). The Cochran-Armitage test of trend assessed the overall trend of response across the dose groups (from the lowest dose [or placebo], to the highest dose); Test type: Other; p = 0.1664, Cochran-Armitage test of trend

2. Secondary Outcome: Percentage of Subjects With New HO at Weeks 6 and 12
Description: Low dose CT scan was used as a secondary imaging assessment of HO and was performed at the same time points as plain radiographs. The percentage of subjects with new HO (regardless of the amount of new HO) at the flare-up site as assessed by CT scan and/or plain radiographs at Weeks 6 and 12 were analysed. The results are from Global Read reviews. The holistic Global Read process allowed concurrent review of all modalities across all time points, and provided access to selected clinical data at the time of review.
Time Frame: Weeks 6 and 12 (Day 84)
Population: The PP population included all subjects who were eligible for the FAS population, completed Week 6 study visit with no major protocol deviations with at least 80% compliance with study drug, and had an evaluable radiograph or CT at Week 6 sufficient to allow determination of HO at flare-up site.
Measure: Number; unit: percentage of subjects
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg | Placebo
Number analyzed (Participants) | 20 | 9 | 10
percentage of subjects
  Week 6 | 15.0 | 22.2 | 30.0
  Week 12 | 15.0 | 44.4 | 40.0
Statistical Analysis 1: Comparison: Palovarotene 10/5 mg vs Palovarotene 5/2.5 mg vs Placebo; Week 6: Cochran-Armitage test of trend (one-sided). The Cochran-Armitage test of trend assessed the overall trend of response across the dose groups (from the lowest dose [or placebo], to the highest dose); Test type: Other; p = 0.2335, Cochran-Armitage test of trend
Statistical Analysis 2: Comparison: Palovarotene 10/5 mg vs Palovarotene 5/2.5 mg vs Placebo; Week 12: Cochran-Armitage test of trend (one-sided). The Cochran-Armitage test of trend assessed the overall trend of response across the dose groups (from the lowest dose [or placebo], to the highest dose); Test type: Other; p = 0.0837, Cochran-Armitage test of trend

3. Secondary Outcome: Change From Baseline in Amount (Area) of New HO Formed at the Flare-up Site at Weeks 6 and 12
Description: Interpretation of plain radiographs document the amount (area) of HO on both the AP and lateral radiograph views. The area for each view was a sum of all the new HO at the flare-up location (and thus if there are multiple HO lesions, the area of each lesion was determined and then the total across all lesions were summed to obtain a total new HO). This total new HO sum was used in the analysis of the area of new HO. Results from Primary Read reviews are presented.
Time Frame: Baseline, Weeks 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: square millimeters (mm)
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg | Placebo
Number analyzed (Participants) | 20 | 9 | 10
square millimeters (mm)
  Week 6: number analyzed (Participants) | 20 | 9 | 9
  Week 6 | 0.00 (0.000) | 38.85 (116.542) | 75.89 (176.744)
  Week 12: number analyzed (Participants) | 20 | 9 | 9
  Week 12 | 19.00 (84.955) | 71.22 (213.650) | 621.71 (1287.519)
Statistical Analysis 1: Comparison: Palovarotene 10/5 mg vs Placebo; Week 6: Analysis of area of new HO; Test type: Other; p = 0.6984, Pairwise test; Least square (LS) mean = -86.35, Standard Error of Mean 220.570
Statistical Analysis 2: Comparison: Palovarotene 5/2.5 mg vs Placebo; Week 6: Analysis of area of new HO; Test type: Other; p = 0.8811, Pairwise test; LS mean = -38.07, Standard Error of Mean 252.192
Statistical Analysis 3: Comparison: Palovarotene 10/5 mg vs Placebo; Week 12: Analysis of area of new HO; Test type: Other; p = 0.0017, Pairwise test; LS mean = -764.38, Standard Error of Mean 220.570
Statistical Analysis 4: Comparison: Palovarotene 5/2.5 mg vs Placebo; Week 12: Analysis of area of new HO; Test type: Other; p = 0.0094, Pairwise test; LS mean = -703.43, Standard Error of Mean 252.192

4. Secondary Outcome: Percentage of Responders at Week 12
Description: A responder was defined as a subject with no or minimal new HO at the flare-up site versus baseline as assessed by plain radiographs at Week 12. Minimal new HO is defined as new HO with an HO score <=3 in both the AP and lateral projections (or if one view is non-interpretable or non-evaluable, then the remaining evaluable view is used). The HO score ranges from 0 to 6 where, 0 = no HO and 6 = single contiguous HO with longest dimension >2 diameters of the reference normotopic bone in any projection. The highest HO score from the 2 projections was used. Results from the Primary Read reviews are presented. The Primary Read process included a double-read radiology review paradigm with consensus adjudication. Radiography and CT scans were examined independently by scan type, flare-up region, and imaging time point in order to determine whether radiography would be sufficient to measure new HO formation.
Time Frame: Baseline and Week 12
Population: The PP population included all subjects who were eligible for FAS population, completed Week 6 study visit with no major protocol deviations with at least 80% compliance with study drug, and had an evaluable radiograph or CT at Week 6 sufficient to allow determination of HO at flare-up site. Only subjects with interpretable outcomes were evaluated.
Measure: Number; unit: percentage of subjects
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg | Placebo
Number analyzed (Participants) | 20 | 9 | 9
percentage of subjects | 95.0 | 88.9 | 77.8
Statistical Analysis 1: Comparison: Palovarotene 10/5 mg vs Palovarotene 5/2.5 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.1503, Cochran-Armitage test of trend

5. Secondary Outcome: Change From Baseline in Bone Specific Alkaline Phosphatase at Weeks 2, 4, 6 and 12
Description: Blood and urine samples for analysis of cartilage, bone, angiogenesis, and inflammation biomarkers were collected. Bone specific alkaline phosphatase was analysed as a bone and cartilage biomarker.
Time Frame: Baseline, Weeks 2, 4, 6 and 12
Population: The FAS population included all subjects who received at least 1 dose of study drug and had at least 1 evaluable post-baseline radiograph or CT sufficient to allow determination of HO at the flare-up site.
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg | Placebo
Number analyzed (Participants) | 21 | 9 | 10
microgram per liter (mcg/L)
  Week 2: number analyzed (Participants) | 15 | 4 | 6
  Week 2 | -1.33 (13.267) | -3.18 (4.619) | 12.02 (35.263)
  Week 4: number analyzed (Participants) | 15 | 7 | 6
  Week 4 | -1.41 (8.328) | 3.80 (12.072) | 7.53 (10.208)
  Week 6: number analyzed (Participants) | 17 | 7 | 7
  Week 6 | -2.53 (8.157) | 0.74 (3.316) | 6.23 (6.851)
  Week 12: number analyzed (Participants) | 16 | 7 | 7
  Week 12 | 2.49 (5.506) | 0.89 (6.738) | 10.00 (10.091)

6. Secondary Outcome: Change From Baseline in C-Reactive Protein at Weeks 2, 4, 6 and 12
Description: Blood and urine samples for analysis of cartilage, bone, angiogenesis, and inflammation biomarkers were collected. C-reactive protein was analysed as a inflammation biomarker.
Time Frame: Baseline, Weeks 2, 4, 6 and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg | Placebo
Number analyzed (Participants) | 21 | 9 | 10
mg/L
  Week 2: number analyzed (Participants) | 13 | 6 | 5
  Week 2 | 8.62 (28.085) | 0.09 (2.370) | -1.59 (1.909)
  Week 4: number analyzed (Participants) | 15 | 7 | 5
  Week 4 | 1.48 (4.924) | 23.26 (38.311) | 2.34 (3.704)
  Week 6: number analyzed (Participants) | 15 | 7 | 6
  Week 6 | 0.14 (3.419) | 2.70 (7.984) | 1.20 (1.319)
  Week 12: number analyzed (Participants) | 15 | 7 | 6
  Week 12 | 2.82 (11.762) | 1.27 (1.789) | -0.30 (2.951)

7. Secondary Outcome: Change From Baseline in C-Terminal Telopeptide at Weeks 2, 4, 6 and 12
Description: Blood and urine samples for analysis of cartilage, bone, angiogenesis, and inflammation biomarkers were collected. C-terminal telopeptide was analysed as a bone and cartilage biomarker.
Time Frame: Baseline, Weeks 2, 4, 6 and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg | Placebo
Number analyzed (Participants) | 21 | 9 | 10
mcg/L
  Week 2: number analyzed (Participants) | 15 | 5 | 5
  Week 2 | -0.020 (0.290) | 0.118 (0.359) | 0.071 (0.342)
  Week 4: number analyzed (Participants) | 16 | 8 | 6
  Week 4 | 0.015 (0.337) | 0.095 (0.380) | 0.188 (0.219)
  Week 6: number analyzed (Participants) | 19 | 8 | 8
  Week 6 | 0.105 (0.304) | 0.078 (0.293) | 0.125 (0.351)
  Week 12: number analyzed (Participants) | 18 | 8 | 7
  Week 12 | 0.116 (0.241) | 0.054 (0.285) | 0.126 (0.197)

8. Secondary Outcome: Change From Baseline in Procollagen Type 1 N-Terminal Propeptide at Weeks 2, 4, 6 and 12
Description: Blood and urine samples for analysis of cartilage, bone, angiogenesis, and inflammation biomarkers were collected. Procollagen type 1 N-terminal propeptide was analysed as a bone and cartilage biomarker.
Time Frame: Baseline, Weeks 2, 4, 6 and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg | Placebo
Number analyzed (Participants) | 21 | 9 | 10
mcg/L
  Week 2: number analyzed (Participants) | 14 | 4 | 5
  Week 2 | 53.022 (72.091) | 78.930 (113.443) | 42.058 (77.358)
  Week 4: number analyzed (Participants) | 15 | 8 | 6
  Week 4 | 123.986 (207.513) | 117.476 (169.238) | 194.193 (318.920)
  Week 6: number analyzed (Participants) | 18 | 8 | 6
  Week 6 | 141.304 (206.163) | 147.409 (246.219) | 252.328 (389.359)
  Week 12: number analyzed (Participants) | 17 | 8 | 6
  Week 12 | 120.489 (211.565) | 25.766 (233.860) | 141.367 (213.926)

9. Secondary Outcome: Change From Baseline in Procollagen Type 1 C-Terminal Propeptide Biomarker at Weeks 2, 4, 6 and 12
Description: Blood and urine samples for analysis of cartilage, bone, angiogenesis, and inflammation biomarkers were collected. Procollagen type 1 C-terminal propeptide was analysed as a bone and cartilage biomarker.
Time Frame: Baseline, Weeks 2, 4, 6 and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg | Placebo
Number analyzed (Participants) | 21 | 9 | 10
mcg/L
  Week 2: number analyzed (Participants) | 15 | 5 | 6
  Week 2 | 22.12 (61.976) | 23.26 (11.585) | 82.93 (109.010)
  Week 4: number analyzed (Participants) | 15 | 8 | 7
  Week 4 | 72.16 (98.697) | 76.10 (110.041) | 140.26 (155.036)
  Week 6: number analyzed (Participants) | 18 | 8 | 8
  Week 6 | 73.36 (130.437) | 87.19 (96.451) | 125.31 (110.389)
  Week 12: number analyzed (Participants) | 17 | 8 | 7
  Week 12 | 51.21 (82.901) | 47.30 (112.113) | 96.49 (92.215)

10. Secondary Outcome: Change From Baseline in Amount of Bone Formation (Volume) at Weeks 6 and 12
Description: Low dose CT scan were used as a secondary imaging assessment of HO, and was performed at the same time points as plain radiographs. Interpretation of the CT scan documented the amount (volume) and grade of HO. The independent reviewer scored HO lesions according to the following scale for HO on CT. Grade 1 = fluid attenuation without evidence of calcification at CT, Grade 2 = calcification of soft tissues without evidence of bone formation, Grade 3 = immature bone formation, and Grade 4 = mature bone with cortical differentiation. Volume of new HO was determined according to the following steps: (1) calculate volume of new HO compared to baseline for each reviewer/HO ID, (2) sum the volume of new HO across HO IDs for each reviewer, and (3) average the volume of new HO across reviewers. Results from Primary Read reviews are presented.
Time Frame: Baseline, Weeks 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cubic mm
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg | Placebo
Number analyzed (Participants) | 20 | 9 | 10
cubic mm
  Week 6: number analyzed (Participants) | 19 | 9 | 10
  Week 6 | 2820.53 (11078.233) | 326.58 (979.733) | 11459.42 (29759.691)
  Week 12: number analyzed (Participants) | 17 | 9 | 10
  Week 12 | 3857.95 (11860.978) | 1184.99 (3188.020) | 16181.64 (41643.976)

11. Secondary Outcome: Percentage of Subjects With Soft Tissue Swelling and Cartilage Formation Assessed by Magnetic Resonance Imaging (MRI) or Ultrasound (US) at Weeks 6 and 12
Description: The MRI was utilized to evaluate the presence of soft tissue swelling/edema (and volume of the swelling/edema) and presence of cartilage formation (yes or no). For subjects who could not have an MRI, US was used to assess edema severity for the sub-set of subjects enrolled after this opinion was introduced in a protocol amendment. Imaging film from MRI was assessed by two independent readers. When there was sufficient agreement between the independent readers on volume, both of the independent readings were used for analysis with the volume measurements averaged. When there was insufficient agreement between the independent readers, an adjudication reading was provided and used for analysis. The US was used for soft tissue swelling/edema but not cartilage formation. Percentage calculated as % = 100 x n/N' where N' is the number of subjects with interpretable outcomes. Results from Primary Read reviews are presented.
Time Frame: Weeks 6 and 12
Population: as for outcome 5
Measure: Number; unit: percentage of subjects
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg | Placebo
Number analyzed (Participants) | 21 | 9 | 10
percentage of subjects
  Soft tissue swelling: Week 6: number analyzed (Participants) | 16 | 8 | 9
  Soft tissue swelling: Week 6 | 50.0 | 50.0 | 66.7
  Soft tissue swelling: Week 12: number analyzed (Participants) | 15 | 9 | 9
  Soft tissue swelling: Week 12 | 60.0 | 66.7 | 66.7
  Cartilage formation: Week 6: number analyzed (Participants) | 13 | 3 | 4
  Cartilage formation: Week 6 | 15.4 | 0.0 | 0.0
  Cartilage formation: Week 12: number analyzed (Participants) | 12 | 3 | 5
  Cartilage formation: Week 12 | 8.3 | 0.0 | 0.0

12. Secondary Outcome: Change From Baseline in Percent of Normal Arc of Motion at the Primary Joint (Flare-up Site) at Weeks 6 and 12
Description: Active range of motion, expressed as the percent of normal arc of motion, measurements at the primary joint associated with the flare-up and adjoining joints was assessed by goniometer.
Time Frame: Baseline, Weeks 6 and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent of normal arc of motion
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg | Placebo
Number analyzed (Participants) | 21 | 9 | 10
percent of normal arc of motion
  Week 6: number analyzed (Participants) | 20 | 8 | 10
  Week 6 | -0.40 (9.574) | -1.36 (21.336) | -0.99 (18.951)
  Week 12: number analyzed (Participants) | 20 | 8 | 10
  Week 12 | 0.58 (15.079) | -4.23 (26.791) | -2.31 (18.963)

13. Secondary Outcome: Subject and Investigator Global Assessment of Movement at Weeks 6 and 12
Description: Flare-up movement outcomes were independently assessed by both the subject (or parent of a subject under 8 years of age) and the Investigator at Weeks 6 and 12 by completing the global assessment of movement. The subject/parent completed the global assessment first. Prior to reviewing the subject's assessment, the Investigator completed his/her own assessment of the flare-up outcome. Subjects were assessed how the flare-up affected their movement on a scale ranging 1 to 5 where, 1 = severely worse movement and 5 = better movement compared with study Day 1 (day of first dose of study drug). Investigators were assessed how the flare-up affected the subject's movement on a scale ranging 1 to 5 where, 1 = severely worse movement and 5 = better movement compared with baseline (day of screening physical examination).
Time Frame: Weeks 6 and 12
Population: The FAS population included all subjects who received at least 1 dose of study drug and had at least 1 evaluable post-baseline radiograph or CT sufficient to allow determination of HO at the flare-up site. Only subjects with non-missing values were presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg | Placebo
Number analyzed (Participants) | 21 | 9 | 10
Participants
  Subject Global Assessment: Week 6: number analyzed (Participants) | 9 | 8 | 6
  Subject Global Assessment: Week 6: Score 1 | 0 | 1 | 0
  Subject Global Assessment: Week 6: Score 2 | 1 | 0 | 0
  Subject Global Assessment: Week 6: Score 3 | 0 | 0 | 1
  Subject Global Assessment: Week 6: Score 4 | 2 | 3 | 2
  Subject Global Assessment: Week 6: Score 5 | 6 | 4 | 3
  Subject Global Assessment: Week 12: number analyzed (Participants) | 13 | 9 | 7
  Subject Global Assessment: Week 12: Score 1 | 0 | 1 | 0
  Subject Global Assessment: Week 12: Score 2 | 0 | 1 | 1
  Subject Global Assessment: Week 12: Score 3 | 1 | 0 | 1
  Subject Global Assessment: Week 12: Score 4 | 6 | 2 | 4
  Subject Global Assessment: Week 12: Score 5 | 6 | 5 | 1
  Investigator Global Assessment: Week 6: number analyzed (Participants) | 9 | 8 | 6
  Investigator Global Assessment: Week 6: Score 1 | 1 | 1 | 0
  Investigator Global Assessment: Week 6: Score 2 | 0 | 0 | 1
  Investigator Global Assessment: Week 6: Score 3 | 0 | 0 | 1
  Investigator Global Assessment: Week 6: Score 4 | 3 | 2 | 3
  Investigator Global Assessment: Week 6: Score 5 | 5 | 5 | 1
  Investigator Global Assessment: Week 12: number analyzed (Participants) | 13 | 9 | 7
  Investigator Global Assessment: Week 12: Score 1 | 1 | 1 | 1
  Investigator Global Assessment: Week 12: Score 2 | 0 | 1 | 0
  Investigator Global Assessment: Week 12: Score 3 | 0 | 1 | 0
  Investigator Global Assessment: Week 12: Score 4 | 8 | 2 | 4
  Investigator Global Assessment: Week 12: Score 5 | 4 | 4 | 2

14. Secondary Outcome: Change From Baseline in Flare-Up Pain and Swelling at Weeks 2, 4, 6, 9 and 12
Description: The pain and swelling associated with flare-ups was evaluated using 2 separate numeric rating scales, one for pain and one for swelling. The pain scale ranges from 0 to 10 where, 0 = no pain and 10 = worst pain ever experienced. The swelling scale ranges from 0 to 10 where, 0 = no swelling and 10 = worst swelling ever experienced. The Faces Pain Scale - Revised (FPS-R) was used for children less than 8 years old. The FPS-R ranges from 0 to 10 where, 0 = no pain and 10 = very much pain in two-point increments.
Time Frame: Baseline, Weeks 2, 4, 6, 9 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg | Placebo
Number analyzed (Participants) | 20 | 9 | 10
units on a scale
  Flare-up pain: Week 2 | -2.5 (2.50) | 0.0 (2.40) | -2.0 (1.76)
  Flare-up pain: Week 4 | -3.2 (2.46) | -1.3 (1.58) | -1.9 (3.14)
  Flare-up pain: Week 6 | -3.5 (2.78) | -1.3 (1.58) | -2.4 (2.91)
  Flare-up pain: Week 9: number analyzed (Participants) | 19 | 8 | 10
  Flare-up pain: Week 9 | -3.8 (2.62) | -1.1 (1.64) | -2.1 (1.85)
  Flare-up pain: Week 12 | -3.6 (2.72) | -1.9 (2.42) | -2.2 (2.53)
  Flare-up swelling: Week 2: number analyzed (Participants) | 20 | 7 | 10
  Flare-up swelling: Week 2 | -1.4 (2.76) | -1.3 (2.93) | -2.3 (2.79)
  Flare-up swelling: Week 4: number analyzed (Participants) | 19 | 8 | 10
  Flare-up swelling: Week 4 | -1.7 (3.30) | -1.9 (1.81) | -2.0 (3.30)
  Flare-up swelling: Week 6: number analyzed (Participants) | 20 | 8 | 10
  Flare-up swelling: Week 6 | -2.2 (3.32) | -2.0 (2.45) | -2.6 (3.50)
  Flare-up swelling: Week 9: number analyzed (Participants) | 19 | 7 | 10
  Flare-up swelling: Week 9 | -2.7 (3.32) | -2.3 (2.43) | -1.9 (4.41)
  Flare-up swelling: Week 12: number analyzed (Participants) | 20 | 8 | 10
  Flare-up swelling: Week 12 | -2.1 (3.73) | -2.5 (2.20) | -2.3 (3.16)

15. Secondary Outcome: Percentage of Subjects Who Used Any Assistive Devices and Adaptations for Daily Living at Weeks 6 and 12
Description: Subjects were given a list of FOP assistive devices and adaptations and asked to select those they use for daily living. The FOP assistive devices and adaptations included mobility aids, care attendants, eating tools, personal care tools/aids, bathroom aids and devices, bedroom aids and devices, home adaptations, work environment adaptations, technology adaptations, sports and recreation adaptations, school, and medical therapies for daily living.
Time Frame: Weeks 6 and 12
Population: as for outcome 5
Measure: Number; unit: percentage of subjects
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg | Placebo
Number analyzed (Participants) | 21 | 9 | 10
percentage of subjects
  Week 6: number analyzed (Participants) | 20 | 9 | 10
  Week 6 | 85.0 | 100.0 | 100.0
  Week 12 | 90.5 | 100.0 | 100.0

16. Secondary Outcome: Duration of Active Symptomatic Flare-up
Description: The duration of active symptomatic flare-up was defined as the number of days the subject reported the presence of symptoms in the diary ('Is your flare-up ongoing today?') from Day 1 to study completion at Day 84. The mean number of days of active, symptomatic flare-up is presented for subjects with evaluable diary data.
Time Frame: From Day 1 to Day 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg | Placebo
Number analyzed (Participants) | 17 | 9 | 8
days | 22.1 (20.53) | 44.1 (38.36) | 34.4 (34.15)

17. Secondary Outcome: Change From Baseline in Percentage of Worst Total Score for FOP-Specific Physical Function Questionnaire (FOP-PFQ) at Weeks 2, 4, 6, 9 and 12
Description: The FOP-PFQ consists of 28 questions rated on scales from 1 to 5, with lower scores denoting more difficulty. The adult form of the FOP-PFQ was administered to subjects 15 years of age and older. There are two Pediatric FOP-PFQ (FOP-PFQ-P) forms: a self-completed form for 8 to 14 year-olds and a parent proxy-completed form for 5 to 14 year-olds. For subjects between 8 to 14 years of age, both the self-completed (for 8 to 14 year-olds) and the proxy-completed (for 5 to 14 year olds) forms of the FOP-PFQ-P were administered. However, only the proxy-completed form was used for analysis. Percentage of worst scores ranges from 0% to 100% with 0% = best possible function and 100% = worst possible function. Change from baseline for each time point is presented.
Time Frame: Baseline, Weeks 2, 4, 6, 9 and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg | Placebo
Number analyzed (Participants) | 21 | 9 | 10
units on a scale
  Week 2 | 0.95 (5.484) | 0.31 (3.818) | 2.11 (6.659)
  Week 4: number analyzed (Participants) | 20 | 9 | 10
  Week 4 | 3.42 (7.932) | 2.67 (7.200) | 2.91 (8.427)
  Week 6: number analyzed (Participants) | 21 | 9 | 9
  Week 6 | 3.79 (7.787) | 2.88 (7.550) | 1.75 (5.980)
  Week 9: number analyzed (Participants) | 19 | 8 | 10
  Week 9 | 1.89 (5.432) | -0.52 (7.881) | 4.91 (13.185)
  Week 12: number analyzed (Participants) | 20 | 9 | 10
  Week 12 | 4.22 (7.915) | 1.08 (8.724) | 3.02 (9.587)

18. Secondary Outcome: Change From Baseline in Physical and Mental Health Using Age-Appropriate Forms of the Patient Reported Outcomes Measurement Information System (PROMIS) Global Health Scale at Weeks 2, 4, 6, 9 and 12
Description: The PROMIS Global Health contains 10 questions which are rated on scales from 1 to 5 or 0 to 10. Global physical health scores were calculated as the sum of scores from parameters 3, 6, 7, and 8 and ranges from 4 to 20 where, 4 = worse health and 20 = better health. Global mental health scores were calculated as the sum of scores from parameters 2, 4, 5, and 10 and ranges from 4 to 20 where, 4 = worse health and 20 = better health. For paediatric subjects, the PROMIS was administered as per the adult version. However, there is a single total score for the paediatric PROMIS (as opposed to global physical and global mental health scores as are in the adult version). The total score were converted to a T-score. A T-score of 50 is normal and increments of 10 are +/- 1 standard deviation away from the norm. A T-score <50 indicates worse health, while a T-score >50 indicates better health. The higher values (positive changes) indicate better health.
Time Frame: Baseline, Weeks 2, 4, 6, 9 and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg | Placebo
Number analyzed (Participants) | 21 | 9 | 10
t-score
  Adult-only: Global Physical Health T-Score: Week 2: number analyzed (Participants) | 17 | 5 | 5
  Adult-only: Global Physical Health T-Score: Week 2 | 2.76 (5.308) | 0.00 (1.768) | 5.90 (2.087)
  Adult-only: Global Physical Health T-Score: Week 4: number analyzed (Participants) | 17 | 5 | 5
  Adult-only: Global Physical Health T-Score: Week 4 | 4.66 (6.590) | 2.66 (4.345) | 5.56 (2.904)
  Adult-only: Global Physical Health T-Score: Week 6: number analyzed (Participants) | 17 | 5 | 4
  Adult-only: Global Physical Health T-Score: Week 6 | 4.69 (5.585) | 7.08 (6.591) | 5.73 (2.750)
  Adult-only: Global Physical Health T-Score: Week 9: number analyzed (Participants) | 15 | 4 | 5
  Adult-only: Global Physical Health T-Score: Week 9 | 4.96 (5.489) | 5.58 (3.381) | 4.94 (3.135)
  Adult-only:Global Physical Health T-Score: Week 12: number analyzed (Participants) | 16 | 5 | 5
  Adult-only:Global Physical Health T-Score: Week 12 | 3.97 (6.764) | 4.98 (6.246) | 3.78 (3.883)
  Adult-only: Global Mental Health T-Score: Week 2: number analyzed (Participants) | 17 | 5 | 5
  Adult-only: Global Mental Health T-Score: Week 2 | 3.66 (5.216) | 3.20 (2.024) | 1.98 (3.124)
  Adult-only: Global Mental Health T-Score: Week 4: number analyzed (Participants) | 17 | 5 | 5
  Adult-only: Global Mental Health T-Score: Week 4 | 3.32 (5.066) | 2.28 (2.700) | 7.30 (5.609)
  Adult-only: Global Mental Health T-Score: Week 6: number analyzed (Participants) | 17 | 5 | 5
  Adult-only: Global Mental Health T-Score: Week 6 | 4.15 (6.878) | 2.54 (4.980) | 4.34 (5.850)
  Adult-only: Global Mental Health T-Score: Week 9: number analyzed (Participants) | 15 | 4 | 5
  Adult-only: Global Mental Health T-Score: Week 9 | 4.62 (7.684) | 1.68 (3.641) | 5.38 (5.438)
  Adult-only: Global Mental Health T-Score: Week 12: number analyzed (Participants) | 16 | 5 | 5
  Adult-only: Global Mental Health T-Score: Week 12 | 4.33 (7.527) | 3.10 (4.127) | 1.04 (3.664)
  Paediatric-only: Global Health T-Score: Week 2: number analyzed (Participants) | 3 | 4 | 3
  Paediatric-only: Global Health T-Score: Week 2 | -2.27 (4.278) | 1.05 (2.352) | -1.80 (4.668)
  Paediatric-only: Global Health T-Score: Week 4: number analyzed (Participants) | 3 | 4 | 3
  Paediatric-only: Global Health T-Score: Week 4 | -0.57 (2.499) | 1.43 (6.352) | -6.40 (4.314)
  Paediatric-only: Global Health T-Score: Week 6: number analyzed (Participants) | 3 | 4 | 3
  Paediatric-only: Global Health T-Score: Week 6 | -2.23 (3.499) | 2.80 (4.955) | -3.30 (7.826)
  Paediatric-only: Global Health T-Score: Week 9: number analyzed (Participants) | 3 | 4 | 3
  Paediatric-only: Global Health T-Score: Week 9 | 1.17 (2.021) | 1.83 (1.434) | -3.50 (4.668)
  Paediatric-only: Global Health T-Score: Week 12: number analyzed (Participants) | 3 | 4 | 3
  Paediatric-only: Global Health T-Score: Week 12 | 0.17 (7.572) | -2.13 (2.964) | -6.57 (1.950)

19. Secondary Outcome: Maximum Measured Plasma Concentration (Cmax) of Palovarotene
Description: The Cmax of palovarotene was determined.
Time Frame: Pre-dose and 3, 6, 10, and 24 hours (hrs) post-dose at Week 2, and at Week 4 or 6
Population: The Pharmacokinetic (PK) population included all subjects who had sufficient blood samples collected for valid estimation of PK parameters.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg
Number analyzed (Participants) | 20 | 8
picograms per milliliter (pg/mL)
  Week 2: number analyzed (Participants) | 15 | 5
  Week 2 | 95620.00 (30296.77) | 35620.00 (19882.08)
  Week 4/Week 6: number analyzed (Participants) | 17 | 7
  Week 4/Week 6 | 45505.88 (17061.05) | 18958.57 (9238.62)

20. Secondary Outcome: Minimum Measured Plasma Concentration (Cmin) of Palovarotene
Description: The Cmin of palovarotene was determined.
Time Frame: Pre-dose and 3, 6, 10, and 24 hrs post-dose at Week 2, and at Week 4 or 6
Population: The PK population included all subjects who had sufficient blood samples collected for valid estimation of PK parameters.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg
Number analyzed (Participants) | 20 | 8
pg/mL
  Week 2: number analyzed (Participants) | 15 | 5
  Week 2 | 3128.53 (2358.88) | 1739.40 (963.68)
  Week 4/Week 6: number analyzed (Participants) | 17 | 7
  Week 4/Week 6 | 3879.00 (7042.29) | 614.14 (289.72)

21. Secondary Outcome: Time of Maximum Measured Plasma Concentration (Tmax) of Palovarotene
Description: The Tmax obtained by inspection of palovarotene was determined.
Time Frame: Pre-dose and 3, 6, 10, and 24 hrs post-dose at Week 2, and at Week 4 or 6
Population: as for outcome 20
Measure: Median (Full Range); unit: hr
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg
Number analyzed (Participants) | 20 | 8
hr
  Week 2: number analyzed (Participants) | 15 | 5
  Week 2 | 3.00 [2.83 to 6.03] | 2.77 [2.08 to 5.88]
  Week 4/Week 6: number analyzed (Participants) | 17 | 7
  Week 4/Week 6 | 3.00 [2.75 to 6.00] | 3.00 [3.00 to 6.00]

22. Secondary Outcome: Apparent Terminal Elimination Half-life (t1/2) of Palovarotene
Description: The t1/2 was calculated as ln(2)/ λz. The number of data points included in the regression was determined by visual inspection, but a minimum of three data points in the terminal phase, excluding Cmax, was required to estimate λz.
Time Frame: Pre-dose and 3, 6, 10, and 24 hrs post-dose at Week 2, and at Week 4 or 6
Population: as for outcome 20
Measure: Median (Full Range); unit: hr
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg
Number analyzed (Participants) | 20 | 8
hr
  Week 2: number analyzed (Participants) | 11 | 4
  Week 2 | 4.33 [3.30 to 6.51] | 5.18 [3.29 to 5.94]
  Week 4/Week 6: number analyzed (Participants) | 16 | 4
  Week 4/Week 6 | 4.39 [3.11 to 6.38] | 4.40 [4.13 to 5.11]

23. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve Over the 24-hr Dosing Interval (AUC[0-24hr]) of Palovarotene
Description: The AUC(0-24hr) was calculated using linear trapezoid rule.
Time Frame: Pre-dose and 3, 6, 10, and 24 hrs post-dose at Week 2, and at Week 4 or 6
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg
Number analyzed (Participants) | 20 | 8
hr*pg/mL
  Week 2: number analyzed (Participants) | 13 | 4
  Week 2 | 686308.92 (246797.81) | 350124.65 (181967.49)
  Week 4/Week 6: number analyzed (Participants) | 17 | 7
  Week 4/Week 6 | 311082.39 (128622.73) | 142748.47 (84838.75)

24. Secondary Outcome: Apparent Clearance of Palovarotene (CL/F)
Description: The CL/F was defined as dose/AUC0-24hr.
Time Frame: Pre-dose and 3, 6, 10, and 24 hrs post-dose at Week 2, and at Week 4 or 6
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg
Number analyzed (Participants) | 20 | 8
L/hr
  Week 2: number analyzed (Participants) | 13 | 4
  Week 2 | 15.55 (7.03) | 12.84 (4.07)
  Week 4/Week 6: number analyzed (Participants) | 17 | 7
  Week 4/Week 6 | 17.71 (7.44) | 19.51 (10.66)

ADVERSE EVENTS:
Time Frame: From first dose of study drug (Day 1) up to and including the Week 12 visit, approximately 85 days.
Description: Treatment-emergent adverse events were those with a start date/time after the first dose of study medication. The safety population included all subjects who received at least 1 dose of study drug (placebo or palovarotene).
Arm/Group | Palovarotene 10/5 mg | Palovarotene 5/2.5 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/21 | 1/9 | 1/10
Other Adverse Events (participants affected / at risk) | 21/21 | 9/9 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palovarotene 10/5 mg (N=21) | Palovarotene 5/2.5 mg (N=9) | Placebo (N=10)
Condition aggravated (General disorders) | 2 (2) | 0 (0) | 0 (0) — Any flare-ups reported during the 12-week duration of the study, which were not the flare-up that qualified the subject for the study, were recorded as adverse events.
Myoclonus (Nervous system disorders) | 1 (4) | 0 (0) | 0 (0)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palovarotene 10/5 mg (N=21) | Palovarotene 5/2.5 mg (N=9) | Placebo (N=10)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Condition aggravated (General disorders) | 13 (27) | 2 (2) | 3 (3) — Any flare-ups reported during the 12-week duration of the study, which were not the flare-up that qualified the subject for the study, were recorded as adverse events.
Pyrexia (General disorders) | 1 (2) | 3 (4) | 1 (1)
Application site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 2 (4) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 2 (5) | 0 (0) | 1 (5)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 1 (2)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (3)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Thyroxine free increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Thyroxine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 8 (9) | 1 (1) | 3 (5)
Dizziness (Nervous system disorders) | 1 (2) | 1 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (3) | 2 (5)
Migraine (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 2 (2) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 7 (8) | 5 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (7) | 1 (1) | 2 (2)
Chapped lips (Gastrointestinal disorders) | 5 (6) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 2 (3) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 17 (38) | 5 (5) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 3 (6) | 2 (2) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Dandruff (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (13) | 1 (4) | 6 (14)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 2 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Radiography was less sensitive than CT for detecting new HO. Thus, Global Read data are presented where available using more sensitive CT scans at Week 12 in the PP population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes